CLINICAL TRIAL: NCT04572594
Title: Study on the Molecular Profile and Molecular Signature of Inflammatory Myofibroblastic Tumor
Brief Title: Molecular Profiling and Molecular Labeling of Inflammatory Myofibroblastic Tumor
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Dong sheng Zhang, Chief physician，professor, Sun Yat-sen University
Other Study IDs: Molecular profiling of IMT
Record Dates: First submitted 2020-09-15; First posted 2020-10-01 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Inflammatory Myofibroblatic Tumor
Keywords: IMT; gene; molecular profiling and molecular markers

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tissue wax block
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Inflammatory myofibroblastic tumor: tissue of Inflammatory myofibroblastic tumor lession

SUMMARY:
Gene mutation is a research hotspot in the occurrence of multiple malignant tumors. The somatic gene mutations of many different types of tumors not only help to study the tumorigenesis mechanism and molecular diagnosis, but also can be used as an ideal therapeutic target. Large-scale gene profiling studies performed by humans in various types of epithelial tumors have confirmed some new gene mutations. However, there are few reports on the detection of genes related to inflammatory myofibroblastic tumor, and humans have not yet understood its molecular content. Therefore, it is necessary to further use molecular detection methods to explore the molecular markers of IMT to facilitate its follow-up precise treatment plan.

DETAILED DESCRIPTION:
Inflammatory myofibroblastic tumor（IMT）is a rare clinical mesenchymal tissue-derived tumor, which can occur in almost all organs and soft tissues, and is characterized by low-grade or borderline tumors.

The diagnosis of inflammatory myofibroblastic tumor is mainly based on histopathology and immunohistochemistry. The treatment is resistant to conventional chemotherapy and radiotherapy. The only curative treatment is complete surgical resection. When IMT shows typical cellular structural features in pathology, the diagnosis is relatively simple. However, in the presence of atypical features, the accurate diagnosis of IMT is still a challenge. Therefore, it is necessary to explore a better diagnostic method. Secondly, there is no individualized treatment method for aggressive IMT patients who relapse and metastasize after surgery. At present, gene mutation is a research hotspot in the occurrence of various malignant tumors. The somatic gene mutations of many different types of tumors not only help to study the tumorigenesis mechanism and molecular diagnosis, but also can be used as an ideal therapeutic target. Large-scale gene profiling studies performed by humans in various types of epithelial tumors have confirmed some new gene mutations. However, there are few reports on the detection of inflammatory myofibroblastic tumor, and humans have not yet understood its molecular content. Therefore, it is necessary to further use molecular detection methods to explore the molecular markers of IMT to facilitate its follow-up precise treatment plan.

ELIGIBILITY:
Inclusion Criteria:

1. From December 2009 to July 2019, patients who were pathologically diagnosed with inflammatory myofibroblastic tumor by Sun Yat-sen University Cancer Center；
2. There are related pathological tissue wax blocks in Sun Yat-sen University Cancer Center;
3. Patient clinical and prognosis tracking data are available.

Exclusion Criteria:

The patient who has a clinically detectable second primary malignant tumor.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: From December 2009 to July 2019, the histopathological diagnosis of inflammatory myofibroblastic tumor was confirmed by surgery or puncture at Sun Yat-sen University Cancer Center.
Sampling Method: Probability Sample
Enrollment: 29 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Establishing gene mutation spectrum of patients with inflammatory myofibroblastic tumor | through study completion，an average of 1 year
  We sequenced the genes in tissue samples from patients with inflammatory myofibroblastic tumor, and then analyzed the data to obtain a gene map of this type of tumor, and provide data support for the diagnosis and treatment of the disease.

SECONDARY OUTCOMES:
Exploring molecular markers for inflammatory myofibroblastic tumor | through study completion，an average of 1 year
  We sequenced tissue samples from patients with inflammatory myofibroblastic tumor, and then analyzed the data to explore molecular markers of this type of tumor, and provide assistance in the diagnosis and targeted therapy of the disease.

CONTACTS AND LOCATIONS:
Overall Officials: Dongsheng Zhang, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Cancer center of SunYat-sen University, Guangzhou, Guangdong, China